CLINICAL TRIAL: NCT01542736
Title: Feasibility of Using Concurrent Carboplatin and Reduced Dose Craniospinal Radiation (24Gy) for Metastatic Medulloblastoma, High-Risk Supratentorial PNET and Metastatic PNET
Brief Title: Concurrent Carboplatin and Reduced Dose Craniospinal Radiation for Medulloblastoma and Primitive Neuroectodermal Tumor (PNET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-1151
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Medulloblastoma; High Risk Supratentorial PNET; Metastatic PNET
MeSH Terms: conditions — Medulloblastoma | interventions — Carboplatin; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reduced radiation with concurrent chemotherapy (Experimental): Reduced dose craniospinal radiation with concurrent carboplatin and vincristine administration
  Interventions: Drug: Carboplatin; Drug: Vincristine; Radiation: 24 Gy

INTERVENTIONS:
Drug: Carboplatin — Administered concurrently with craniospinal radiation.
Drug: Vincristine — Administered concurrently with craniospinal radiation.
Radiation: 24 Gy — Craniospinal radiation.

SUMMARY:
The purpose of this study is to study the efficacy of the combination of reduced dose craniospinal radiation (reduced from standard of care dosing at 36 Gy to 24 Gy) with concurrent carboplatin and vincristine administration for metastatic classical histology medulloblastomas and high-risk supratentorial PNETs and metastatic PNETs.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 3 years and less than 25 years
* Patients with classic histology or desmoplastic histology metastatic medulloblastoma by histological diagnosis and by head and spine MRI.
* Patients with high-risk supratentorial, non-metastatic, PNET
* Patients with metastatic PNET
* Newly diagnosed patients who have not received prior therapy, with the exception of one short course of emergent chemotherapy in newly presenting patients with neurological compromise per provider decision
* Only patients who are expected to survive at least 6 weeks will be eligible for this study.

Exclusion Criteria:

* Patients who are pregnant may not be treated on this study
* Patients with anaplastic histology

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Madden, RN, CPNP, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reduced Radiation With Concurrent Chemotherapy
Started | 8
Completed | 7
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Reduced Radiation With Concurrent Chemotherapy
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 8.125 [3 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: MRIs of the head and spine. Number of participants with event free survival at 60 months is reported.
Time Frame: Up to 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Radiation With Concurrent Chemotherapy
Number analyzed (Participants) | 8
Participants | 7

2. Primary Outcome: Overall Survival
Description: Overall Survival will be measured at the end of study. number of surviving participants is reported.
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Radiation With Concurrent Chemotherapy
Number analyzed (Participants) | 8
Participants | 7

3. Primary Outcome: Intellectual Competence Measured by IQ Score: Week 8
Description: Neuropsychological testing will be performed after radiation in completed. The Wechsler Intelligence Scale for Children, 5th edition (WISC-V) measures intellectual competence in Verbal Comprehension, Visual Spatial, Fluid Reasoning, Working Memory, and Processing Speed. The average score for the scale is fixed at 100, with a standard deviation of 15. Higher scores indicate higher levels of intellectual competence and a better outcome.
Time Frame: Week 8
Population: Not all participants were feeling well enough to complete testing at this timepoint.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Reduced Radiation With Concurrent Chemotherapy
Number analyzed (Participants) | 5
score on a scale | 102.4 [84 to 122]

4. Primary Outcome: Intellectual Competence Measured by IQ Score: Month 24
Description: Neuropsychological testing will be performed after radiation in completed. IQ score is reported. The Wechsler Intelligence Scale for Children, 5th edition (WISC-V) measures intellectual competence in Verbal Comprehension, Visual Spatial, Fluid Reasoning, Working Memory, and Processing Speed. The average score for the scale is fixed at 100, with a standard deviation of 15. Higher scores indicate higher levels of intellectual competence and a better outcome.
Time Frame: Month 24
Population: Not all participants were feeling well enough to complete testing at this timepoint.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Reduced Radiation With Concurrent Chemotherapy
Number analyzed (Participants) | 6
score on a scale | 96.83 [80 to 127]

5. Primary Outcome: Intellectual Competence Measured by IQ Score: Month 60
Description: as for outcome 4
Time Frame: Month 60
Population: Not all participants were feeling well enough to complete testing at this timepoint.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Reduced Radiation With Concurrent Chemotherapy
Number analyzed (Participants) | 2
score on a scale | 79 [75 to 83]

ADVERSE EVENTS:
Time Frame: Until time of death or progression (Up to 10 years)
Arm/Group | Reduced Radiation With Concurrent Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Radiation With Concurrent Chemotherapy (N=8)
Death due to multi-system organ failure (Infections and infestations) | 1 (1) — Death was related to infection and occurred off-treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Radiation With Concurrent Chemotherapy (N=8)
Relapse (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-08-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT01542736/Prot_000.pdf